CLINICAL TRIAL: NCT04988204
Title: Pilot Study: Diabetes Prevention Program for the Treatment of Nonalcoholic Fatty Liver Disease
Brief Title: Diabetes Prevention Program for the Treatment of Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Amreen Dinani, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 18-1283
Record Dates: First submitted 2021-07-28; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Patients enrolled in 1 year program
  Interventions: Behavioral: Diabetes Prevention Program

INTERVENTIONS:
Behavioral: Diabetes Prevention Program — The Diabetes Prevention Program is a 1 year validated program to prevent the development of type 2 diabetes. Participants with NAFLD will engage will work with a CDC certified DPP certified lifestyle coach and other participants in a group setting during the study focusing on lifestyle changes to achieve weight loss and improvement in NAFLD.

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a rapidly growing epidemic worldwide and is an increasingly important etiology of chronic liver disease and hepatocellular carcinoma. NAFLD affects approximately 90 million people in the United States (US) amounting to an annual cost of $100 billion yearly. It is projected to become the leading cause of liver transplantation in the US by 2030 and is associated with significant morbidity and mortality. NAFLD is a spectrum of liver diseases, ranging from simple steatosis (nonalcoholic fatty liver, NAFL) to hepatic steatosis associated with inflammation (nonalcoholic steatohepatitis, NASH), which can be associated with liver scarring (hepatic fibrosis) and cirrhosis. There are limited therapeutic options that have been shown to effectively reduce or reverse the progression of disease.

Lifestyle modification is the backbone of therapy, but difficult to achieve. A modest amount of weight loss of approximately 3% can reduce liver steatosis and a 10% weight loss can reduce the NASH and improve liver fibrosis. The American Association of the Study of Liver Diseases (AASLD) guidelines state that "a combination of a hypocaloric diet (daily reduction by 500-1000 kcal) and moderate intensity exercise is the best likelihood of sustaining weight loss over time." There are several barriers to adopting a healthy lifestyle involving both patient and physician limitations. The aim of this study is to engage patients in a lifestyle intervention program that has already been shown to be successful in achieving weight loss goals and adopting healthier lifestyle patterns.

The CDC Diabetes Prevention Program, (DPP) was a large (n=3,234) multicenter study aimed to evaluate the effect of lifestyle intervention or treatment with metformin on the incidence of type 2 diabetes (T2DM). Lifestyle intervention reduced the incidence of T2DM by 58% (95% CI, 48-66%) and metformin reduced the incidence by 31% (95% CI, 17-43%) as compared to placebo. To prevent one case of diabetes over three years, 6.9 persons would have to participate in the lifestyle-intervention program, and 13.9 would have to receive metformin. The CDC DPP program has been adapted and tested in the multiple different community and state-wide programs including the YMCA, WorkWellNYC and NYS DPP. In these real-world models, the life style intervention program has been delivered in a group-based format by DPP lifestyle coaches. These programs have been successful like that of the randomized trial and improvements were sustainable at 6 and 12 month follow up after completion of the program. The program is now available and reimbursable through Medicare (Medicare Diabetes Prevention Program).

In this pilot study, the researchers will enroll 20 patients with NAFLD in an adapted DPP program and follow study participants for 1 year. The rationale for the proposed research is to apply the DPP to NAFLD because of the close relationship with Diabetes and determine the real-world outcome of the DPP program on weight loss in patients with NAFLD. If the researchers illustrate that weight loss can be achieved and is sustainable in patients with NAFLD enrolled in lifestyle intervention programs, the researchers can develop innovative approaches to deliver such a program nationwide in a cost-effective and sustainable manner.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of NAFLD, defined by the presence of hepatic steatosis with vibration controlled transient elastography (VCTE) controlled attenuation parameter (CAP) measurement over 240dB/m, or liver biopsy showing macrovesicular steatosis in ≥ 5% of hepatocytes.
* patients were 18 years and older,
* fluent in English (the program could only be conducted in English by the DPP-certified coach),
* able to meet program scheduling requirements, and able to participate in physical activity.

Exclusion Criteria:

* additional causes of liver disease such as viral hepatitis, biliary obstruction, hepatocellular carcinoma, Wilson's disease, Budd Chiari Syndrome, autoimmune hepatitis, alcoholic liver disease or alcohol use (>20g/day women, >30g/day men),
* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values >300 U/L,
* using steatogenic medications (amiodarone, methotrexate, tamoxifen, and corticosteroids),
* pregnant,
* a history of liver transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Number of participants in the program at the end of the study | 12 months
  Retention defined as number of patients in the program at the end of the study

SECONDARY OUTCOMES:
Change in Weight | baseline and 12 months
  Change in Weight at 12 months as compared to baseline
Hepatic steatosis via Fibroscan | Baseline
  Changes in hepatic steatosis measured with fibroscan using the controlled attenuated parameter.
Hepatic steatosis via Fibroscan | 6 months
  Changes in hepatic steatosis measured with fibroscan using the controlled attenuated parameter .
Hepatic steatosis via Fibroscan | 12 months
  Changes in hepatic steatosis measured with fibroscan using the controlled attenuated parameter.
Glycosylated A1C | Baseline
  Glycosylated A1C in assessing metabolic comorbidity
Glycosylated A1C | 6 months
  Glycosylated A1C in assessing metabolic comorbidity
Glycosylated A1C | 12 months
  Glycosylated A1C in assessing metabolic comorbidity
Lipid levels | Baseline
  Lipid levels in assessing metabolic comorbidity
Lipid levels | 6 months
  Lipid levels in assessing metabolic comorbidity
Lipid levels | 12 months
  Lipid levels in assessing metabolic comorbidity
Liver enzymes levels | Baseline
  Liver enzymes levels for ALT, AST, and ALP
Liver enzymes levels | 6 months
  Liver enzymes levels for ALT, AST, and ALP
Liver enzymes levels | 12 months
  Liver enzymes levels for ALT, AST, and ALP
Bilirubin level | Baseline
  Liver enzyme level for Bilirubin
Bilirubin level | 6 months
  Liver enzyme level for Bilirubin
Bilirubin level | 12 months
  Liver enzyme level for Bilirubin

CONTACTS AND LOCATIONS:
Overall Officials: Amreen Dinani, Principal Investigator — Icahn School of Medicine, Division of Liver Diseases
Locations (1):
- Mount Sinai Union Square, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
was not including inn protocol and consent form

REFERENCES:
- [Derived] Hershman M, Torbjornsen K, Pang D, Wyatt B, Dieterich DT, Perumalswami PV, Branch AD, Dinani AM. Modification of the diabetes prevention program for the treatment of nonalcoholic fatty liver disease: A pilot study. Obes Sci Pract. 2022 Oct 20;9(3):218-225. doi: 10.1002/osp4.637. eCollection 2023 Jun. PMID 37287520